CLINICAL TRIAL: NCT06837480
Title: Placebo-Controlled Phase II Randomized Clinical Trial of Photobiomodulation Therapy in Head and Neck Cancer Survivors With Chronic Lymphedema
Brief Title: Photobiomodulation in Head and Neck Cancer-Related Chronic Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jie Deng, Professor, PhD, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UPCC 01325; Pending (Other: National Cancer Institute)
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Lymphedema of the Head and Neck
Keywords: Head and neck cancer, chronic lymphedema, photobiomodulation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- ARM A: PBMT12 (Active Comparator): After completion of the baseline measures, participants in ARM A will be scheduled for PBMT twice a week for 6 weeks followed by sham therapy once per week for 6 weeks (a total of 18 sessions: 12 PBMT and 6 sham therapy sessions).
  Interventions: Device: LTU-904 Portable Laser Therapy Unit (active laser device); Device: LTU-904 Portable Laser Therapy Unit (sham/inactive laser device)
- ARM B: PBMT18 (Active Comparator): After completion of the baseline measures, participants in ARM B will be scheduled for PBMT twice a week for 6 weeks followed by PBMT once per week for 6 weeks (a total of 18 PBMT sessions).
  Interventions: Device: LTU-904 Portable Laser Therapy Unit (active laser device)
- ARM C: Placebo (Sham Comparator): After completion of the baseline measures, participants in ARM C will receive sham therapy, twice a week for 6 weeks followed by sham therapy once per week for 6 weeks (a total of 18 sham therapy sessions).
  Interventions: Device: LTU-904 Portable Laser Therapy Unit (sham/inactive laser device)

INTERVENTIONS:
Device: LTU-904 Portable Laser Therapy Unit (active laser device) — The RianCorp LTU-904 laser therapy unit (active laser device) will be used for photobiomodulation therapy (PBMT).
  Arms: ARM A: PBMT12; ARM B: PBMT18
Device: LTU-904 Portable Laser Therapy Unit (sham/inactive laser device) — The RianCorp LTU-904 laser therapy (sham/inactive laser device) unit will be used for sham therapy.
  Arms: ARM A: PBMT12; ARM C: Placebo

SUMMARY:
The U.S. Food and Drug Administration approved photobiomodulation therapy (PBMT) as a treatment for breast cancer-related arm lymphedema (BCRL) in 2006. The investigators conducted two pilot clinical trials. Results demonstrated the feasibility, acceptability, and preliminary efficacy of PBMT for the treatment of chronic lymphedema in head and neck cancer (HNC) survivors. The objective of this study is to further investigate and confirm the positive effects of PBMT on HNC-related chronic lymphedema.

ELIGIBILITY:
Inclusion Criteria:

>18 years of age Biopsy proven head and neck cancer No evidence of cancer at the time of study enrollment, between 12- and 60-month post-cancer treatment Chronic lymphedema (defined as lymphedema persisting for a minimum of 6 months) A minimum of 2 sites of external lymphedema At least 1 site with lymphedema of moderate severity as assessed using the HN-LEF Assessment Criteria Failed lymphedema therapy (defined as any of the following: incomplete response to therapy, progression of lymphedema after therapy, inability to perform effective self-care resulting in fluid re-accumulation; and inability to complete treatment due to systems barriers). In addition, patients must be able to understand English in order to complete questionnaires; and to provide informed consent.

Exclusion Criteria:

Patients will be excluded if they have any of the following medical conditions that would prohibit the safe implementation of PBMT:

Women of childbearing age and potential Acute cellulitis within the soft tissues in the head and neck region Chronic inflammatory diseases Venous thrombosis Carotid artery stenosis Requiring ongoing use of diuretics and corticosteroids Pre-existing skin rash, ulceration, open wound in the treatment area Active lymphedema or physical therapy (including hyperbaric oxygen or trental) Allergic and other systemic skin diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Total Severity of External Lymphedema | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Head and Neck Lymphedema and Fibrosis Assessment Criteria.
  External lymphedema is measured by HN-LEF Assessment Criteria. The total external lymphedema severity score is calculated by summing the severity score of each site (total 9 sites, severity score ranging from 0-27). For each site, the severity of LEF includes no lymphedema (=0), mild (=1), moderate (=2), and severe (=3).
  Change in total severity of external lymphedema from baseline to 12-month post-intervention visits. A larger reduction in this score means more reduction in the severity of external lymphedema.

SECONDARY OUTCOMES:
Total Severity of Internal Lymphedema | Pre-intervention, after 18 sessions (end-of-intervention), 12-month post-intervention
  Modified Patterson Scale
  Endoscopic exams were performed by a trained oncology provider. Internal lymphedema was scored using the Modified Patterson Scale, which documents internal swelling in the oral cavity, pharynx, and larynx. Four grades are used to rate edema level (normal = 0, mild = 1, moderate = 2, and severe = 3) for each anatomical structure. Sites are marked "N/A" when they are unable to be evaluated. The scale has good intra-rater reliability (weighted kappa, 0.84) and moderate inter-rater reliability (weighted kappa, 0.54).
  Change in total severity of external lymphedema from baseline to 12-month post-intervention visits. A larger reduction in this score means more reduction in the severity of external lymphedema.
Symptom Burden Score | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Head and Neck Lymphedema and Fibrosis Symptom Inventory
  Symptom burden is assessed by Head and Neck Lymphedema and Fibrosis Symptom Inventory (HN-LEF SI). Higher scores (score ranging from 0-5) indicate increased symptom burden.
  Change in symptom burden score from baseline to 12-month post-intervention. A larger reduction in this score means decreased symptom burden.
Jaw Range of Motion Degree | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Jaw Range of Motion Scale
  Jaw Range of Motion Scale is a validated scale with a ruler in millimeters to measure mouth opening.
  Change in jaw range of motion degree from baseline to 12-month post-intervention. A larger increase in this degree means better outcome with increased jaw range of motion.
Neck Range of Motion Degree | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Cervical Range of Motion Scale
  Cervical Range of Motion Device, a valid and reliable tool, will be used to measure the amount of neck movement (degrees) for the following neck movements: forward flexion, extension, right and left lateral flexion, and right and left rotation.
  Change in neck range of motion degree from baseline to 12-month post-intervention. A larger change in this degree means better outcome with increased neck range of motion.
Shoulder Range of Motion Degree | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Goniometry
  Goniometry is a validated and reliable tool for measuring shoulder range of motion.
  Change in shoulder range of motion degree from baseline to 12-month post-intervention. A larger change in this degree means better outcome with increased shoulder range of motion.
Quality of Life Score | Pre-intervention, after 12 sessions, after 18 sessions (end-of-intervention), 3-, 6-, 9-and 12-month post-intervention
  Quality of Life Scale (Linear Analog Self-Assessment, LASA)
  Quality of Life Scale (Linear Analog Self-Assessment, LASA) has been extensively used in cancer (e.g., HNC) patients. The scale has shown good reliability (alpha=.83-.88) and good concurrent/construct validity. It covers four major components of QOL (i.e., physical, emotional, spiritual, and intellectual).
  Change in quality of life score from baseline to 12-month post-intervention. A larger increase in this score means better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No